CLINICAL TRIAL: NCT05202366
Title: An Open-label Cosmetic Study to Evaluate the Effectiveness of CGB-400 Topical Gel for Improving Appearance of Toenails Affected by Fungal Infection
Brief Title: An Open-label Study Evaluating the Effectiveness of CGB-400 Topical Gel for Fungal Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CAGE Bio Inc. (Industry)
Collaborators: John Peter Smith Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CGB-405
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Fungal Infection; Onychomycosis; Tinea Unguium
Keywords: Fungal growth; Fungal infection; Onychomycosis; Nail trauma
MeSH Terms: conditions — Mycoses; Onychomycosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Only one treatment group (CGB-400 Topical Gel) will be used for analysis
  Interventions: Drug: CGB-400 Topical Gel

INTERVENTIONS:
Drug: CGB-400 Topical Gel — CGB-400 Gel contains two main ingredients: geranic acid and choline. Geranic acid, a naturally occurring essential oil/terpenoid, is a key ingredient in lemon grass and is also found in other natural materials such as cardamom. The other main ingredient in CAGE is choline, which is an essential dietary component and found in foods as free choline and as several esterified forms such as phosphocholine and phosphatidylcholine.
  Other Names: CGB-400C Gel

SUMMARY:
The goal of the current study is to evaluate the ability of CGB-400, a proprietary eutectic mixture of GRAS compounds, to clear the toenail fungal growth and improve the appearance of the fungus affected area(s).

This is an open-label, single group POC study evaluating the effectiveness of CGB-400 Topical Gel for toenail fungal growth clearing. The study consists of a 12-week period with 5 clinic visits at the following timepoints: Baseline (Day 0), and Weeks 2, 6, and 12 and post-application follow-up at Week 24. The applications could be extended for an additional 12 weeks based on PI's observations.

Approximately 15 subjects will be enrolled and subjected to application of CGB-400 Topical Gel. Subjects must be at least 18 years of age and will be selected by the concerned PI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 (and ≤99) at the time of Informed Consent.
2. Nail fungal infection of at least one great toe [per visual assessment by the clinical investigator]
3. Subjects who have target toenail showing 20-65% involvement as judged by the clinical investigator.
4. Subject must be physically able to reach toes to clean them and apply product.
5. Subject is willing to discontinue use of other nail fungus treatment products and nail cosmetic products for duration of this study.
6. Subject is willing and available to return for study follow up.
7. Signed written informed consent form (ICF) prior to any trial related activity (subjects must have the mental, literate, and legal ability to give a written informed consent, which must comply with the ICH GCP guidelines and local requirements.
8. Agree to take and share pictures of the treated toenails on a periodic basis during the study and follow-up period.

Exclusion Criteria:

1. Female subjects that are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
2. Known hypersensitivity or previous allergic reaction to any constituent of the Investigational Product (i.e., essential oils, fragrance, choline, phosphatidylcholine, propylene glycol, limonene, cellulose).
3. Nails with clinical evidence of no or low distal growth.
4. History or presence of another skin/nail condition/disease that is located in the treatment area(s) and might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, psoriasis, significant actinic damage, vitiligo, open wounds, infection, etc.).
5. Basal cell carcinoma within 6 months of Visit 1.
6. Uncontrolled systemic disease.
7. Foreseen unprotected and intense/excessive UV exposure during the course of the study.
8. Use of prohibited concomitant medications/procedures, as specified below in Table 2, during the study or within the defined washout periods.
9. Scheduled or planned surgical procedures during the course of the study.
10. Unable or unwilling to comply with any of the study requirements.
11. Medical or psychiatric conditions, or a personal situation, that may increase the risk associated with study participation or may interfere with interpretation of study results or subject compliance and, in the opinion of the PI, makes the subject inappropriate for study entry.
12. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
13. Exposure to any other investigational drug/device within 30 days prior to study entry.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female ≥18 (and ≤99) at the time of Informed Consent will be involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) of affected toenails | 24 weeks
  Clear 0% nail involvement
  1. Almost clear 0%-≤10% nail involvement
  2. Mild 10%-<25% nail involvement
  3. Moderate 25%-≤50% nail involvement
  4. Severe >50%-≤75% nail involvement

SECONDARY OUTCOMES:
Percent clear area on affected toenail/region (s) | 24 weeks
  *Clear nail is defined as area from proximal nail fold till most proximal area of abnormality with evidence of persistent clear growth.
  Clearance must be progressively observed over two time points.
Visual inspection (pictures to be collected) | 24 weeks
  Visual inspection for application site reactions: performed at each visit along with images taken by subjects and at the time of clinic visit

OTHER OUTCOMES:
Subject Global Assessment | 24 weeks
  The Subject Global Assessment will be collected in the form "subject questionnaire"
  SUBJECT QUESTIONNAIRE:
  The Investigator (or designate) will ask the following questions at the Baseline visit and subject's answers will be recorded:
  1. How frequently do you typically experience fungal growth each month?
  2. How do you rate your fungal growth today relative to other times?
  3. Are you aware of specific triggers that aggravate fungal growth?
  4. How do you deal with or treat fungal growth?
  5. What other products have you tried in the past for managing/treating fungal growth?
  6. Are there any other aspects of fungal growth or experience that we should know about?

CONTACTS AND LOCATIONS:
Overall Officials: Travis Motley, DPM, Principal Investigator — JPS
Locations (1):
- John Peter Smith Hospital, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 24 weeks
Access Criteria: Research data, in hard copy or electronic form (CDs, DVDs, digital or magnetic tape, hard-drives, flash-memory drives, etc.) will be stored and managed in a secure manner following federal guidelines and according to state and institutional policies and practices. Further, research documents including electronic documents containing subject data, identifiers and linked data will be securely stored in locked containers (file cabinets, lockers, drawers, etc.) in accordance with standard document management practices. At all times, only listed key personnel specifically designated and authorized by the Principal Investigator shall have access to any research related documents. All such personnel will be properly trained and supervised regarding the management and handling of confidential materials. The Principal Investigator assumes full responsibility for such training, supervision, and conduct.